CLINICAL TRIAL: NCT05357989
Title: A 6-month Prospective, Randomized, Double-blind, Placebo-controlled Clinical Trial Investigating the Efficacy, Safety, and Tolerability of Two Different Doses of Buntanetap or Placebo in Patients With Early Parkinson's Disease
Brief Title: A Double-blind Study to Investigate Efficacy and Safety of Buntanetap Compared With Placebo in Participants With Early PD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Annovis Bio Inc. (Industry)
Collaborators: TFS Trial Form Support (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ANVS-22001
Record Dates: First submitted 2022-04-19; First posted 2022-05-03 (Actual); Results first posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Parkinson's Disease, Idiopathic
Keywords: Parkinson's
MeSH Terms: conditions — Parkinson Disease | interventions — phenserine

STUDY DESIGN:
Intervention Model Description: Randomized
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 10 mg buntanetap/posiphen (Experimental): Buntanetap/posiphen 10 mg oral capsule with daily administration for a period of 6 months
  Interventions: Drug: buntanetap/posiphen
- 20 mg buntanetap/posiphen (Experimental): Buntanetap/posiphen 20 mg oral capsule with daily administration for a period of 6 months
  Interventions: Drug: buntanetap/posiphen
- Placebo (Placebo Comparator): Placebo oral capsule with daily administration for a period of 6 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: buntanetap/posiphen — HPMC (vegetarian source) capsule shells
  Other Names: Posiphen Tartrate; ANVS401
  Arms: 10 mg buntanetap/posiphen; 20 mg buntanetap/posiphen
Drug: Placebo — HPMC (vegetarian source) capsule shells
  Arms: Placebo

SUMMARY:
The purpose of this study is to measure safety and efficacy of buntanetap/posiphen capsules compared with placebo capsules in participants with early PD.

Study details include:

* The study duration will be up to 7-8 months.
* The double-blind treatment duration will be up to 6 months.
* There will be 5 in-clinic visits and 7 phone calls

DETAILED DESCRIPTION:
450 early Parkinson's Disease (PD) patients will be randomized to 10mg, 20 mg of buntanetap/posiphen or placebo. They will undergo a Screening Visit, and if they provide informed consent and are considered eligible per the inclusion and exclusion criteria, will proceed to participate in the treatment period. Randomized participants will visit the clinic for the first-time dosing in clinic with administration of 10 mg or 20mg of buntanetap/posiphen or placebo, followed by an at home dosing period of 6 months, with daily administration of 10 mg or 20mg of buntanetap/posiphen or Placebo. Participants will be required to visit clinics 1 month, 2 months, 3 months, and 6 months (end-of-trial), where they will undergo study procedures that include safety assessments (AE and concomitant medication monitoring, 12-lead ECGs, clinical laboratory testing, vital signs assessments, and physical examinations) and psychometric tests (MDS-United Parkinson's Disease Rating Scale (MDS-UPDRS), Clinical Global Impression of Severity (CGIS), Wechsler Adult Intelligence Scales (WAIS), Mini-Mental State Examination (MMSE)) and Participant Global Impression of Change (PGIC). At the end of blood sampling, the subjects will need to stay for a minimum of 1 hour of observation. After all end-of-study procedures are complete, the subject will be discharged to home. A 24-hour follow-up call will occur after all clinical visits to assess the participants current condition and if there are any additional adverse events to report.

Buntanetap/posiphen has shown to improve PD subjects' mobility. MDS-UPDRS sum of score of Part II + Part III and Total score of all four parts will be measured to assess its improvement on PD subjects daily living, mobility and complications. PGIC will also be measured to assess its effect.

Buntanetap/posiphen has shown to reduce inflammation and preserve axonal integrity and synaptic functions as well as neurotoxic proteins in previous Phase 2a studies. In this study we plan to measure plasma glial fibrillary acidic protein (GFAP), neurofilament light (NFL) and potentially TDP43.

Reports of adverse events (AEs) and serious adverse events (SAEs) during exposure to buntanetap/posiphen will be collected to evaluate if there are any significant clinical safety issues for the study population. Extensive clinical and laboratory safety data already exist for buntanetap/posiphen; therefore, these safety measures will be sufficient in the proposed study.

For clinical, functional, and cognitive assessment measures, The subjects will be administered the Hoehn & Yahr and the MMSE for determination of inclusion into the study. The MDS-UPDRS and PGIC will be administered for subjects' movement and daily function. The Coding subtest from the WAIS 4th edition will serve as a sensitive measure of Central Nervous System (CNS) dysfunction. MMSE will also be measured to assess subjects' cognitive change.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of idiopathic Parkinson Disease according to MDS Clinical Diagnostic Criteria for Parkinson's Disease.
2. H&Y score =1, 2 or 3 during ON-state & OFF-state <2hrs per day.
3. Male or female aged 40 - 85 years.
4. MMSE score between the range of 22-30 during screening visit (ON-state) and subjects can live independently without a caregiver.
5. Female subjects of childbearing potential* must have a negative serum or urine pregnancy test at Screening, must be non-lactating and must agree to use a highly effective method of contraception (i.e., a method resulting in a failure rate of less than 1% per year when used consistently and correctly) during the trial and for 4 weeks after the last dose of trial treatment, such as:

   * Oral, intravaginal, or transdermal combined (estrogen plus progestogen) hormonal contraception associated with inhibition of ovulation
   * Oral, injectable, or implantable progestogen-only hormonal contraception associated with inhibition of ovulation
   * Intrauterine device (IUD)
   * Intrauterine hormone-releasing system (IUS)
   * Bilateral tubal occlusion
   * Vasectomized partner (a vasectomized partner is a highly effective contraception method provided that the partner is the sole male sexual partner of the participant, and the absence of sperm has been confirmed. If not, an additional highly effective method of contraception should be used)
   * Sexual abstinence (sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatment. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the study and the preferred and usual lifestyle of the participant) *Non-childbearing potential includes surgically sterilized or postmenopausal with no menstrual bleeding for at least one year prior to study start.
6. Male subjects must be sterile or sexually inactive or agree not to father a child during the study and one month after the last dose of study medication and must agree to use a barrier method for contraception. Female partners of male subject must adopt a highly effective method of contraception with a failure rate of less than 1% per year when used consistently and correctly such as:

   * Oral, intravaginal, or transdermal combined (estrogen plus progestogen) hormonal contraception associated with inhibition of ovulation
   * Oral, injectable, or implantable progestogen-only hormonal contraception associated with inhibition of ovulation
   * Intrauterine device (IUD)
   * Intrauterine hormone-releasing system (IUS)
   * Bilateral tubal occlusion 6. Female participants will be given a urine pregnancy test at the screening visit for which they should test negative.
7. General cognition and functional performance sufficiently preserved that the subject can provide written informed consent.
8. No evidence of current suicidal ideation or previous suicide attempt in the past month as evaluated in the Columbia Suicide Severity Rating Scale.
9. Stability of permitted medications prior to screening for at least 4 weeks.
10. At screening subjects do not need to but may be on the following medication:

    * Standard of Care anti-parkinsonian medication
    * Anticonvulsant medications used for epilepsy or mood stabilization, neuropathic pain indications
    * Mood-stabilizing psychotropic agents, including, but not limited to, lithium.
11. Adequate visual and hearing ability (physical ability to perform all the study assessments).
12. Good general health with no disease expected to interfere with the study.
13. Subjects previously exposed to buntanetap can still be included in the study after a 28- day wash out period.

Exclusion Criteria:

1. Has a history of a psychiatric disorder such as schizophrenia, bipolar disorder or major depression according to the criteria of the most current version of the Diagnostic and Statistical Manual of Mental Disorders (DSM). Mild depression or history of depression that is stable on treatment with a selective serotonin reuptake inhibitor (SSRI) or selective norepinephrine reuptake inhibitor (SNRI) medication at a stable dose is acceptable.
2. History of a seizure disorder, if stable on medication is acceptable.
3. Has a history or current evidence of long QT syndrome, Fridericia's formula corrected QT (QTcF) interval ≥ 475ms, or torsades de pointes.
4. Has bradycardia (<50 bpm) or tachycardia (>100 bpm) on the ECG at screening.
5. Has uncontrolled Type-1 or Type-2 diabetes. A subject with HbA1c levels up to 7.5% can be enrolled if the investigator believes the subject's diabetes is under control.
6. Has clinically significant renal or hepatic impairment.
7. Has any clinically significant abnormal laboratory values. Subjects with liver function tests (aspartate aminotransferase [AST] or alanine aminotransferase [ALT]) greater than twice the upper limit of normal will be excluded.
8. Is at imminent risk of self-harm, based on clinical interview and responses on the C SSRS, or of harm to others in the opinion of the Investigators. Subjects must be excluded if they report suicidal ideation with intent, with or without a plan or method (e. g. positive response to Items 4 or 5 in assessment of suicidal ideation on the C SSRS) in the past 2 months, or suicidal behavior in the past 6 months.
9. Has cancer or has had a malignant tumor within the past year, except subjects who underwent potentially curative therapy with no evidence of recurrence. (Subjects with stable untreated prostate cancer or skin cancers are not excluded).
10. Alcohol / Substance use disorder, moderate to severe, in the last 5 years according to the most current version DSM.
11. Participation in another clinical trial with an investigational agent and have taken at least one dose of study medication, unless unblinded on placebo, within 60 days prior to the start of screening. The end of a previous investigational trial is the date the last dose of an investigational agent was taken, or five half-lives of the investigational drug, whichever is greater.
12. Subjects with learning disability or developmental delay.
13. Subjects whom the site PI deems to be otherwise ineligible.
14. Subjects with a known allergy to the investigational drug or any of its components.
15. Subject is currently pregnant, breast-feeding and/or lactating.
16. Subject is currently taking CYP3A4 inhibitors and/or inducers.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 523 (Actual)
Dates: Start 2022-08-03 (Actual); Primary Completion 2023-12-04 (Actual); Study Completion 2023-12-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (69):
- United States (43):
  - University of Alabama at Birmingham (UAB)- The Kirklin Clinic, Birmingham, Alabama
  - Banner Sun Health Research Institute - Cleo Roberts Center for Clinical Research, Sun City, Arizona
  - Parkinson's & Movement Disorder Institue (PMDI) - Orange County Office, Fountain Valley, California
  - UCSF Medical Center - Parkinson's Disease and Movement Disorders Clinic, San Francisco, California
  - Rocky Mountain Movement Disorder Center, Englewood, Colorado
  - Ki Health Partners LLC D/B/A New England Institute for Clinical Research, Stamford, Connecticut
  - Visionary Investigators Network, Aventura, Florida
  - Parkinson's Disease and Movement Disorders Center of Boca Raton, Boca Raton, Florida
  - The Neurology Institute - Coral Springs, Coral Springs, Florida
  - Arrow Clinical trial, Daytona Beach, Florida
  - Accel Research Sites - DeLand Clinical Research Unit, DeLand, Florida
  - Coral Clinic Reserach LLC, Homestead, Florida
  - Homestead Associates in Research, Inc, Miami, Florida
  - Visionary Investigators Networks, Miami, Florida
  - Medical Professional Clinical Research Center, INC, Miami, Florida
  - Reliant Medical Research, Miami, Florida
  - Ezy Medical Research Co., Miami, Florida
  - Visionary Investigators Network, Miami, Florida
  - Renstar Medical Research, Ocala, Florida
  - Visionary Investigators Network, Pembroke Pines, Florida
  - Parkinsons Disease Treatment Center, Port Charlotte, Florida
  - University of South Florida (USF) - University of South Florida College of Medicine- Parkinson's Disease and Movement Disorders Center, Tampa, Florida
  - ClinCloud, LLC, Viera, Florida
  - Conquest Research, LLC, Winter Park, Florida
  - CenExel iResearch, LLC, Decatur, Georgia
  - Hawaii Pacific Neuroscience, LLC, Honolulu, Hawaii
  - Josephson Wallack Munshower Neurology, P.C., Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - Michigan State University (MSU)- Health Team- Neurology and Ophthalmology Clinic, East Lansing, Michigan
  - Quest Research Institue, Farmington Hills, Michigan
  - Parkinson's Disease and Movement Disorders Center of Long Island, Commack, New York
  - Mount Sinai West (Mount Sinai Roosevelt), New York, New York
  - Ohio State University Wexner Medical Center (OSUWMC) - CarePoint Gahanna, Columbus, Ohio
  - The Movement Disorder Clinic (MDC) of Oklahoma, Tulsa, Oklahoma
  - Abington Neurology, Abington, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina (MUSC) - The Murray Center for Research on Parkinson's Disease and Related Disorders, Charleston, South Carolina
  - Veracity Neuroscience, LLC, Memphis, Tennessee
  - Central Texas Neurology Consultants, Round Rock, Texas
  - University of Virginia Health System (UVAHS)- Adult Neurology Clinic, Charlottesville, Virginia
  - Inland Northwest Research, Spokane, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Germany (7):
  - Curiositas-ad-sanum GmbH, Haag, Bavaria
  - Kliniken Beelitz GmbH - Neurologisches Frachkrankenhaus fur Bewegungsstoerungen / Parkinson, Beelitz, Brandenburg
  - Paracelsus-Kliniken Deutschland GmbH & Co. KGaA - Paracelsus-Elena-Klinik Kassel, Kassel, Hesse
  - University Hospital Muenster, Münster, North Rhine-Westphalia
  - Klinik und Poliklinik fur Neurologie - Universitatsklinikum Carl Gustav Carus an der Techischen Universitat, Dresden, Saxony
  - Neurologie Berlin - Gemeinschaftspraxis Dr. Ehret / Dr. von Pannwitz, Berlin
  - Alexianer St. Joseph-Krankenhaus Berlin-Weissensee, Berlin
- Hungary (2):
  - Debreceni Egyetem Klinikai Központ Neurológiai Klinika (Kenézy Gyula Campus, Neurológiai Osztály), Debrecen
  - PTE AOK Neurologiai Klinika, Pécs
- Italy (3):
  - Universita degli Studi di Salerno - Centro per le Malattie Neurodegenerative, Baronissi, Campania
  - San Raffaele Cassino - Centro di Cura e Prevenzione per il Parkinson, Cassino, Lazio
  - San Raffaele Pisana - Centro per la Cura e la Diagnosi del Parkinson, Rome, Lazio
- Poland (7):
  - Pratia MCM Krakow, Krakow, Lesser Poland Voivodeship
  - Unicardia Specjalstyczne Centrum Leczenia Chorob Serca I Naczyn&Unimedica Specjalistyczne Centrum Medyczne, Krakow, Lesser Poland Voivodeship
  - Krakowska Akademia Neurologil Sp. z o.o. - Centrum Neurologii Klinicznej, Krakow, Lesser Poland Voivodeship
  - RCMed Oddzial Sochaczew, Sochaczew, Masovian Voivodeship
  - MTZ Clinical Research Powered by Pratia, Warsaw, Masovian Voivodeship
  - Specjalistyczna Praktyka Lekarska Dr. Stanislaw Ochudlo, Katowice, Silesian Voivodeship
  - NEURO-CARE Sp. z o.o. Sp. Komandytowa, Siemianowice Śląskie, Silesian Voivodeship
- Spain (7):
  - Hospital General Universitario de Elche, Elche, Alicante
  - Hospital Universitaris General de Catalunya (HGC), Sant Cugat del Vallès, Barcelona
  - Policlinica Gipuzkoa - Centro de Invesigacion Parkinson (CIP), Donostia / San Sebastian, Gipuzkoa
  - Universidad Complutense de Madrid (UCM) - Hospital Universitario Infanta Sofia, San Sebastián de los Reyes, Madrid
  - Universidad de Navarra - Clnica Universidad de Navarra (CUN) - Pamplona, Pamplona, Navarre
  - Universidad de Navarra - Clinica Universidad de Navarra (CUN) - Madrid, Madrid
  - Hospital Universitario Virgen del Rocio (URVR - Instituto de Biomedicina de Sevilla (IBIS), Seville

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | 10 mg Buntanetap/Posiphen | 20 mg Buntanetap/Posiphen
Started | 176 | 174 | 173
Completed | 162 | 159 | 150
Not Completed | 14 | 15 | 23

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 10 mg Buntanetap/Posiphen | 20 mg Buntanetap/Posiphen | Total
Number analyzed (Participants) | 176 | 174 | 173 | 523
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.4 (8.88) | 65.0 (8.85) | 65.4 (10.09) | 65.2 (9.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 54 | 55 | 174
  Male | 111 | 120 | 118 | 349
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 30 | 21 | 31 | 82
  Not Hispanic or Latino | 146 | 152 | 141 | 439
  Unknown or Not Reported | 0 | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 4 | 4 | 3 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 6 | 3 | 13
  White | 167 | 163 | 166 | 496
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 1 | 0 | 0 | 1
Mini-Mental State Examination (MMSE) [Mean (Standard Deviation); unit: units on a scale] — Population: Not all participants completed the MMSE at Baseline.
  units on a scale
    number analyzed (Participants) | 173 | 173 | 171 | 517
    (all) | 28.7 (1.71) | 28.7 (1.70) | 28.3 (2.12) | 28.6 (1.86)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Month 6 in MDS-UPDRS Part II (OFF-state)
Description: Change in the Score from the MDS- Unified Parkinson's Disease Rating Scale (UPDRS) Parts II from Baseline to the End of Trial. MDS-UPDRS Part II (Motor experiences of daily living) has 13 items and the score ranges from 0-52, with higher scores reflecting greater severity.
Time Frame: Baseline and 6 months visits
Population: Participants with MDS-UPDRS Part II scores at Baseline and 6 months (intent-to-treat population)
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 10 mg Buntanetap/Posiphen | 20 mg Buntanetap/Posiphen
Number analyzed (Participants) | 160 | 160 | 152
units on a scale | -0.10 (0.311) | 0.57 (0.312) | -0.04 (0.319)

2. Secondary Outcome: Change From Baseline to Month 6 in the MDS-UPDRS Part III (OFF-state)
Description: MDS-UPDRS Part III (motor examination) has 18 items and ranges from 0-132, with higher scores reflecting greater severity.
Time Frame: Baseline and 6 months visits
Population: Participants with MDS-UPDRS Part III scores at Baseline and 6 months (intent-to-treat population)
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 10 mg Buntanetap/Posiphen | 20 mg Buntanetap/Posiphen
Number analyzed (Participants) | 160 | 160 | 153
units on a scale | -2.90 (0.698) | -1.04 (0.697) | -2.66 (0.713)

3. Other Pre Specified Outcome: Change From Baseline to Month 6 in MMSE (OFF-state)
Description: Change in the MMSE score from Baseline to the End of Trial. MMSE is a brief screening instrument used to assess cognitive function (orientation, memory, attention, ability to name objects, follow verbal/written commands, write a sentence, and copy figures). Total score ranges from 0 to 30 with a lower score indicating greater disease severity.
Time Frame: Baseline and 6 months visits
Population: Participants with MMSE scores at Baseline and 6 months (intent-to-treat population)
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 10 mg Buntanetap/Posiphen | 20 mg Buntanetap/Posiphen
Number analyzed (Participants) | 159 | 159 | 152
units on a scale | -0.39 (0.123) | -0.08 (0.123) | -0.05 (0.126)

4. Post Hoc Outcome: Change From Baseline to Month 6 in MMSE (OFF-state) for Participants With Baseline MMSE Scores 20-28
Description: as for outcome 3
Time Frame: Baseline and 6 months visits
Population: Participants with MMSE scores at Baseline and 6 months
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 10 mg Buntanetap/Posiphen | 20 mg Buntanetap/Posiphen
Number analyzed (Participants) | 49 | 50 | 54
units on a scale | -0.50 (0.317) | 0.65 (0.313) | 0.45 (0.301)

ADVERSE EVENTS:
Time Frame: From consent to end of trial (up to 8 months)
Arm/Group | Placebo | 10 mg Buntanetap/Posiphen | 20 mg Buntanetap/Posiphen
All-Cause Mortality (participants affected / at risk) | 0/176 | 1/174 | 0/173
Serious Adverse Events (participants affected / at risk) | 5/176 | 4/174 | 11/173
Other Adverse Events (participants affected / at risk) | 20/176 | 15/174 | 24/173
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=176) | 10 mg Buntanetap/Posiphen (N=174) | 20 mg Buntanetap/Posiphen (N=173)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Angina Pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Myocardial Ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Accidental Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Hip Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Toxic Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Addison's Disease (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis Acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=176) | 10 mg Buntanetap/Posiphen (N=174) | 20 mg Buntanetap/Posiphen (N=173)
Covid-19 (Infections and infestations) | 10 (10) | 5 (5) | 4 (4)
Nausea (Gastrointestinal disorders) | 5 (5) | 5 (5) | 11 (14)
Fatigue (General disorders) | 5 (5) | 5 (6) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Annovis Bio's agreements with its investigators may vary. However, Annovis Bio does not prohibit any investigator from publishing. Any publications from a single site are postponed until the publication of the pooled data for a clinical trial or for 12 months.

DOCUMENTS (2):
  • Study Protocol (2023-08-21): https://cdn.clinicaltrials.gov/large-docs/89/NCT05357989/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-11): https://cdn.clinicaltrials.gov/large-docs/89/NCT05357989/SAP_001.pdf